CLINICAL TRIAL: NCT02987894
Title: Prospective Observation of Aortic Regurgitation After TAVI and Progress Over Time: PROGRESS PVL Registry
Acronym: PROGRESS
Status: Completed | Type: Observational
Sponsor: Symetis SA (Industry)
Responsible Party: Sponsor
Organization: Boston Scientific Corporation (Industry)
Other Study IDs: 2016-02
Record Dates: First submitted 2016-10-27; First posted 2016-12-09 (Estimated); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Aortic Stenosis
Keywords: TAVI; Transcatheter Aortic Valve Replacement; Transcatheter Aortic Valve Implant; Transfemoral access; Aortic valve regurgitation
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: ACURATE neo™ Aortic Bioprosthesis — TAVI, transcatheter aortic valve replacement. Transfemoral access.
  Other Names: ACURATE TF™ Transfemoral Delivery System

SUMMARY:
The purpose of this post-market registry is to collect and monitor ongoing safety and performance clinical data of the ACURATE neo™ Aortic Bioprosthesis, and the ACURATE TF™ Transferral Delivery System, when used as per IFU.

DETAILED DESCRIPTION:
The primary objective of this post-market registry is to further evaluate the safety and performance of the ACURATE neo™ Aortic Bioprosthesis and the ACURATE TF™ Transferral Delivery System in 500 consented patients with severe aortic stenosis and treated according to the instructions for use (IFU).

Examinations to evaluate the aortic valve regurgitation performed as standard of care in patients undergoing transcatheter aortic valve replacement will be analyzed by an external Core Laboratory. These examinations are limited to echocardiography and/or contrast aortography assessments.

The secondary objective is to collect adverse events and evaluate them according to the VARC-2 consensus document.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is included in the registry if eligible for transcatheter treatment of severe aortic stenosis with the ACURATE neo™ Aortic Bioprosthesis and ACURATE TF™ Transfemoral Delivery System as per the Instructions for Use (Patients which are included but treated outside of the approved indication will be followed for safety reasons).
2. Patient is willing to participate in the study, provides signed Informed Consent/Data Authorization Form and authorizes the sharing of data in the registry. Patient agrees that anonymized imaging data will be sent to and analyzed by an external Core Laboratory.
3. The treating physician should ensure the subject will return for all required post procedure follow-up visits.

Exclusion Criteria:

1. Patients are excluded from the registry if they are not eligible for transcatheter treatment of severe aortic stenosis with the ACURATE neo™ Aortic Bioprosthesis and ACURATE TF™ Transfemoral Delivery System as per the Instructions For Use.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All patients eligible for transcatheter treatment of severe aortic stenosis with the ACURATE neo™ Aortic Bioprosthesis and ACURATE TF™ Transfemoral Delivery System according to the indication in the Instruction for Use.
  The ACURATE neo™ Aortic Bioprosthesis and its Delivery System are indicated for use in patients 75 years of age and older with severe aortic stenosis (mean aortic gradient > 40 mmHg or peak jet velocity > 4.0 m/s or aortic valve area < 1.0 cm2) for whom conventional surgical aortic valve replacement is considered high risk for mortality or who are not operable as determined either by a heart team consisting of a cardiologist and surgeon or by the following risk assessments:
  Logistic EuroSCORE > 20%
  STS score > 10%
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2017-01-02 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Change in total aortic regurgitation over time. | post-implantation on index procedure date, 7- days post-index procedure / discharge (whichever occurs first), 30 days post-index procedure and 12 months post-index procedure
  total aortic regurgitation post procedure, at 7 days or discharge, 30 days and 12 months follow-up

SECONDARY OUTCOMES:
Incidence of all-cause mortality | 30 days post-index procedure
  Incidence of all-cause mortality at 30 days post index procedure
Clinical events as defined per VARC-2 consensus document (VARC-2) | Procedure, 7 days post-index procedure / discharge (whichever occurs first), 30 days post-index procedure and 12 months post-index procedure
  Clinical events as defined per VARC-2 consensus document
Number of patients with procedural success according to VARC II criteria | at index- Procedure
  Procedural success is defined as
  Absence of intra-procedure mortality and complications arising during implantation of the prosthetic valve such as:
  * inability to properly seat the valve in the annulus
  * need for more than one implanted aortic bioprosthesis (valve-in-valve or ectopic deployment)
  * surgical aortic valve replacement required to correct a severe aortic regurgitation or procedure complication The procedure can be considered as success despite the presence of residual aortic regurgitation which may be due to the anatomic configuration of the annulus or a calcific valvular annulus.
Number of patients with device success | 7-days post-index procedure or discharge (whichever occurs first)
  Device success is defined as:
  * Absence of intra-procedure mortality (procedure to 24H) AND,
  * Correct positioning (placement in the annulus with no impairment of aortic bioprosthesis function) of a single prosthetic heart valve into the proper anatomical location AND,
  * Intended performance of the prosthetic heart valve:
    * No prosthesis-patient mismatch (EAOi >0.85 cm2/m2) AND,
    * Mean aortic valve gradient <20mmHg or peak velocity < 3 m/s AND,
    * No moderate or severe prosthetic valve regurgitation.
  In evaluating echo parameters, values at 7D/Discharge (whichever occurs first) will be used for each of the echo parameters above. If any of echo parameters is missing at 7-days or discharge, post-procedure data may be used for the missing values. If device success or failure cannot be determined due to missing of parameters listed above or un-evaluable echocardiography assessment, device success will be considered not obtainable.
Number of patients with adverse events assessed by VARC-2 Composite Safety | 30 days post-index procedure
  VARC-2 Composite Safety at 30 days defined as:
  * All-cause mortality
  * All stroke (disabling and non-disabling)
  * Life-threatening bleeding
  * Acute kidney injury - Stage 2 or 3 (including renal replacement therapy)
  * Coronary artery obstruction requiring intervention
  * Major vascular complication
  * Valve-related dysfunction requiring repeat procedure (BAV, TAVI or SAVI)
Functional improvement | 7 days post-index procedure or discharge (whichever occurs first), 30 days post-index procedure and 12 months post-index procedure
  Functional improvement from baseline as per NYHA Functional Classification
Hemodynamic function improvement from baseline | 7 days post-index procedure or discharge (whichever occurs first), 30 days post-index procedure and 12 months post-index procedure
  Improvement from baseline of the hemodynamic function: effective orifice area and mean transprosthetic gradient
Valve related dysfunction | 7 days post-index procedure or discharge (whichever occurs first), 30 days post-index procedure and 12 months post-index procedure
  Valve related dysfunction defined as: mean aortic valve gradient ≥ 20mmHg, EOA ≤0.9-1.1 cm2, and/or DVI< 0.35, and/or moderate or severe prosthetic valve regurgitation (See VARC-2 and Figure 4 from VARC manuscript)

CONTACTS AND LOCATIONS:
Overall Officials: Won-Keun Kim, Dr, Principal Investigator — Kerckhoff-Klinik Forschungsgesellschaft mbH
Locations (23):
- Canada (2):
  - London Health Sciences Centre, University Hospital, London, Ontario
  - Saint Paul's Hospital, Porvidence Health Care Institute, Vancouver
- Germany (17):
  - Klinikum Augsburg, Augsburg
  - Zentralklinik Bad Berka, Bad Berka
  - Kerkhoff Kilnik, Bad Nauheim
  - Immanuel Hospital Bernau- Herzzentrum Brandenburg, Bernau
  - Universitätsklinikum, Cologne
  - Sana-Herzzentrum Cottbus GmbH, Cottbus
  - St Johannes Hospital, Dortmund
  - Goethe Universität, Frankfurt
  - Universitätklinikum Giessen, Giessen
  - Universitätsklinikum Halle, Halle
  - Universitätsklinikum Jena, Jena
  - Städisches Klinikum Karlsruhe GmbH, Karlsruhe
  - Helios Klinik Fur Herzzchirurgie Karlsruhe, Karlsruhe
  - Sana Herzzentrum Leipzig, Leipzig
  - Universitätsklinikum Münster, Münster
  - Städische Kliniken, Neuss
  - Universitätsklinikum Tübingen, Tübingen
- Italy (2):
  - Ospedale Civile di Legnano, Legnano
  - Fondazione Toscana G.Monasterio, Ospedale del Cuore G.Pasquinucci, Massa
- United Kingdom (2):
  - University Hospital NHS, Leicester
  - Oford University Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Undecided
The data and study protocol for this clinical trial may be made available to other researchers in accordance with the Boston Scientific Data Sharing Policy (http://www.bostonscientific.com/en-US/data-sharing-requests.html).